CLINICAL TRIAL: NCT02728986
Title: Comparative and Prospective Evaluation of Direct Cost of Venous Leg Ulcers Management With Two Compression Systems
Brief Title: Cost Evaluation of Venous Leg Ulcers Management
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FR Study No-05-000001; 2014-A01128-39 (Other: ANSM)
Record Dates: First submitted 2016-03-29; First posted 2016-04-06 (Estimated); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Varicose Ulcer
Keywords: Costs and Cost Analysis; Humans; Health Care Costs; varicose ulcer; Compression Bandages
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Compression1 (Active Comparator): Multilayer compression bandage (Profore)
  Interventions: Device: Profore
- Compression2 (Experimental): Coban2 compression system
  Interventions: Device: Coban2

INTERVENTIONS:
Device: Profore — Profore multilayer compression bandage + standard regimen for wound care according to investigator's choice
  Arms: Compression1
Device: Coban2 — Coban2 compression system + standard regimen for wound care according to investigator's choice
  Arms: Compression2

SUMMARY:
The purpose of this study is to evaluate direct costs of Venous Leg Ulcers (VLU) management when two different compression systems are used.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate direct costs of Venous Leg Ulcers management when two different compression systems are used. Micro-costing during the study will bring direct costs which include nurse and physician time, dressings and bandages.

Perspective of costs will be Public Health Insurance. Time horizon will be 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* consent to participate
* ambulatory management
* 1 to 3 leg ulcers
* leg ulcers below the knee and above ankle
* no contra-indication to wear compression bandage
* not currently treated by one of the investigational devices

Exclusion Criteria:

* cognitive impairment
* opposition to wear compression bandage
* bedridden
* pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2015-12-17 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Direct cost of leg ulcer management | 16 weeks
  Direct cost includes cost of bandages, dressings, nurse/doctor visits. Cost will be computed upon consumptions reported by healthcare professionals.

SECONDARY OUTCOMES:
Prevalence of adverse events related to compression | 16 weeks
  Number and type of adverse events related to compression bandages
Patient's compression bandage acceptance score | 16 weeks
  Four ad hoc 7-level Likert scales will be used to assess bandage impact on daily activities, sleep, shoes and slippage
Number of patients with fully healed ulcer | 16 weeks
  Full healing rate
EuroQoL 5D-5L change between baseline and last visit | 16 weeks
  Quality of Life
Average time to full healing | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Meaume, MD, Study Chair — AP-HP Hôpital Rothschild - Paris
Locations (1):
- Quimper Center, Quimper, France

IPD SHARING:
Plan to Share IPD: Undecided